CLINICAL TRIAL: NCT01350765
Title: Naushero Feroze Neonatal Survival Project: A Cluster Randomized Trial to Determine the Effectiveness of Package of Community Based Interventions to Reduce Neonatal Deaths Due to Birth Asphyxia, Low Birth Weight & Neonatal Sepsis
Brief Title: Naushero Feroze Neonatal Survival Project
Acronym: AKU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Save the Children (Other); Pakistan Ministry of Health (Other Government)
Responsible Party: Principal Investigator, Dr Zulfiqar Ahmed Bhutta, Professor and Founding Chair, Division of Women and Child Health, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1212-Ped/ERC
Record Dates: First submitted 2011-05-09; First posted 2011-05-10 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Birth Asphyxia; Very Low Birth Weight Baby; Neonatal Sepsis
Keywords: Birth asphyxia; Low birth weight; neonatal sepsis; mortality; community based interventions
MeSH Terms: conditions — Asphyxia Neonatorum; Neonatal Sepsis | interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): This would be the interventional arm of the study, where the LHWs would receive additional training for identification and management of birth asphyxia, lbw, and sepsis.
  Interventions: Behavioral: Intervention
- Control (Active Comparator): This would be the comparative group of the study in which the LHWs would perform the usual routine tasks assigned to them by their program.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Intervention — The LHWs of the selected intervention areas would receive additional training on ENC for identification, management and referral for birth asphyxia, lbw and neonatal sepsis.
  Arms: Intervention
Behavioral: Control — The LHWs in the control areas would perform their routine tasks as assigned to them by their program
  Arms: Control

SUMMARY:
The present study will be carried out in close collaboration with the National Program for Lady Health Workers, a Ministry of Health program with 100,000 Lady Health Workers covering 60% of the rural population of Pakistan. A team of Lady Health Workers and a Traditional Birth Attendant will provide care to the mothers and newborns at household level. A Basic Health Unit will take care of non complicated referrals and provide injectable antibiotics for neonatal sepsis. Complicated (definitions given in methods section) cases will be referred by the LHWs/BHUs to the District Headquarter Hospital which will have a functioning neonatal care unit. The District Health Services, Naushero Feroz, Provincial Department of Health, Sindh and the Federal Ministry of Health are study collaborators, therefore, guaranteeing scaling up of interventions at national level.

Hypothesis:

In comparison to a basic package of existing training program of LHWs, enhanced training of LHWs and TBAs in the early recognition and management of birth asphyxia, serious newborn infections and LBW (combined with prompt referral) will result in an additional 30% reduction in neonatal mortality.

DETAILED DESCRIPTION:
The proposed body of work addresses important major determinants and immediate causes of neonatal mortality in Pakistan. The recent DHS survey indicates that three causes prematurity, birth asphyxia and serious infections account for approximately 85% of the burden of newborn deaths in Pakistan (PDHS 2007). The recent evidence base of interventions for neonatal interventions clearly indicates that the investigators have a basis for action and several interventions that can make a difference to outcomes. Several of these interventions are clearly feasible within the health system and a fundamental point would be the assurance of skilled care and services for newborn resuscitation, basic preterm care and management of referred cases with neonatal infections within the health facilities (RHCs, THQ and DHQ hospitals in the catchment district). However, given the fact that the vast majority of neonatal birth and deaths still occur in community settings, the added value is the implementation of relevant interventions in community settings. To illustrate, the figure below indicates the potential interventions, links between them and pathways for reduction in the exposure to and adverse outcomes from neonatal sepsis. Although the algorithm suggests that severe neonatal infections should be referred for further care in facility settings, it is recognized that in some situations where care seeking may neither be possible nor feasible, treatment for neonatal sepsis may need to be provided at domiciliary or community level (i.e. through community based clinics or BHUs).

Research questions

Can a package of community-based interventions, linked to strengthened health facilities, reduce NMR and be feasibly delivered, with interventions focused on training TBAs & LHWs to be linked such that LHWs recognize and provide immediate/early management of the newborn complications - birth asphyxia, serious newborn infection, and low birth weight, in tandem with TBAs?

Can these community-based cadres of care providers improve and sustain skills for the provision of quality care for newborn complications of birth asphyxia, serious newborn infection, and low birth weight?

Can community-based strategies of training TBAs and LHWs, and mobilizing communities to focus on perinatal health, result in improved knowledge and use of key newborn health practices related to prevention of newborn complications such as birth asphyxia, serious newborn infections, and complications low birth weight?

Primary Objectives:

To develop and implement intervention packages for TBAs and LHWs to reduce the burden of birth asphyxia, sepsis and low birth weight and asses their feasibility for potential scale up

To assess the efficacy of this intervention package in reducing all cause neonatal mortality at population level

Secondary Objectives:

To improve case recognition and management of birth asphyxia, sepsis and LBW by primary care health care providers (in both the public and private sector such as Midwives, LHWs and TBAs) in primary care settings.

To evaluate the combined effectiveness of birth asphyxia, sepsis and low birth weight interventions delivered by TBAs and LHWs on cause specific neonatal mortality at population level.

To evaluate the effectiveness of using the enhanced intervention package to enhance collaboration and linkages between LHWs and TBAs and to increase LHW attendance during home deliveries.

ELIGIBILITY:
Inclusion Criteria:

Children of ages 1 day to 28 days, within the catchment area of the preformed research.

Exclusion Criteria:

Those who are not willing to participate in the study.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 37201 (Actual)
Dates: Start 2010-03; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
neonatal mortality rate Perinatal mortality rates Neonatal mortality rates | two year
  the subjects from the two arms would be inquired on information pertaining to socioeconomic position, health services, behaviors and morbibity/ mortality. in view of the most reported concern in the previous studies is noenatal mortality, that information will be primarily important for this research.

SECONDARY OUTCOMES:
Cause specific mortality rates (due to birth asphyxia,neonatal sepsis and low birth weight) | two years

CONTACTS AND LOCATIONS:
Overall Officials: Sajid B Soofi, MBBS, FCPS, Study Director — Aga Khan University; Zulfiqar A Bhutta, PhD, Principal Investigator — Aga Khan University
Locations (1):
- Pediatric Resaerch Office, Naushahro Fīroz, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes